CLINICAL TRIAL: NCT00014911
Title: Islet Transplantation for Type 1 Diabetic Patients Using the Edmonton Protocol of Steroid Free Immunosuppression (ITN005CT)
Brief Title: Islet Transplantation for Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN005CT (DAIT NIS01)
Record Dates: First submitted 2001-04-13; First posted 2001-08-31 (Estimated); Results first posted 2012-10-17 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation; Sirolimus; Tacrolimus; Daclizumab; Sulfamethoxazole; Ganciclovir; Trimethoprim; Pentamidine

ARMS (1):
- Islet Transplantation (Experimental): All study participants
  Interventions: Procedure: Islet Transplantation; Drug: Sirolimus; Drug: Tacrolimus; Drug: Daclizumab; Drug: Sulfamethoxazole; Drug: Ganciclovir; Drug: Trimethoprim; Drug: Pentamidine

INTERVENTIONS:
Procedure: Islet Transplantation — Participants will receive portal vein islet infusions (up to 3), e.g., islet transplantations, with a targeted total of exceeding 10,000 islet equivalents per kilogram of body weight (IE/kg) per infusion. Up to three transplants are possible depending on individual results.
Drug: Sirolimus — Administered at a dose of 0.2 mg/kg by mouth once pre-transplantation then 0.1 mg/kg daily post-transplantation. Dosing will be adjusted to achieve a trough peripheral blood level of 12-15 ng/mL x3 months after transplantation and 7-12 ng/mL for the remainder of the study.
Drug: Tacrolimus — Administered at a dose of 1 mg by mouth once pre-transplantation followed by 1 mg twice daily post transplantation. Levels will be adjusted to achieve a peripheral blood trough level of 3-6 ng/mL for maintenance immunosuppression.
Drug: Daclizumab — Administered at a dose of 1 mg/kg intravenously immediately pre-transplantation and 2, 4, 6, and 8 weeks post-transplantation, totaling 5 doses(over 8 weeks). Further daclizumab dosing may be necessary based on individual results and islet transplantation needs.
Drug: Sulfamethoxazole — An antibacterial used to prevent opportunistic infections
Drug: Ganciclovir — An antiviral used to kill viruses and stop viral replication
Drug: Trimethoprim — An antibacterial used to prevent opportunistic infections
Drug: Pentamidine — An antiprotozoal used to prevent disease

SUMMARY:
The purpose of this study is to test whether the islet cell transplantation procedures and results from a previous study in Edmonton, Canada, can be repeated. The study also is designed to learn more about diabetes control using islet cell transplantation.

This is a Phase I/II study (a study that examines effectiveness and looks for side effects). The transplanting of islet cells has been studied in Type 1 diabetic patients whose blood sugar levels will not stay normal, despite intensive insulin therapy. A recent study conducted in Edmonton, Canada, was able to demonstrate that islet transplantation led to insulin independence in a majority of the patients treated. This study extends the results obtained from the Edmonton study, which used islet transplantation in Type 1 diabetic patients with steroid-free immunosuppression.

DETAILED DESCRIPTION:
This is a Phase I/II study (a study that examines effectiveness and looks for side effects). The transplanting of islet cells has been studied in Type 1 diabetic patients whose blood sugar levels will not stay normal, despite intensive insulin therapy. A recent study conducted in Edmonton, Canada, was able to demonstrate that islet transplantation led to insulin independence in a majority of the patients treated. This study extends the results obtained from the Edmonton study, which used islet transplantation in Type 1 diabetic patients with steroid-free immunosuppression.

Eligible patients were randomly selected from the total pool of people who applied through the Immune Tolerance Network. Patients will receive at least 10,000 "islet equivalents" per kilogram (2.2 pounds) of body weight. This likely will require 2 separate islet infusions from 2 separate donors. Immediately before the first transplant, patients will be given anti-rejection (immune suppressing) drugs, including tacrolimus and sirolimus (orally) and daclizumab (intravenously). The islets will be infused into the liver through a tube placed in the portal vein. Heparin (a medication to prevent blood clots) will be administered with the islet infusion. A longer-acting form of heparin will also be given by daily injections during the next week after each transplant. After surgery, patients will receive insulin intravenously for 24 hours. Patients will have an abdominal ultrasound and blood tests to determine liver function. If fewer than 10,000 islets were transplanted, patients will continue insulin treatment, with the dosages adjusted if necessary to account for the transplanted islets. They will take daclizumab every 2 weeks for 8 weeks and tacrolimus and sirolimus daily. Patients will be given antibiotics to prevent infections. Blood tests to determine how much immunosuppressant drug is in the blood will be performed until the drug is at a stable level. Periodically there will be tests to see if the islet cells are functioning. Blood will be drawn to check drug levels and for other tests routinely. Daily insulin requirements will be checked, and these will be recorded monthly. Patients will be followed for at least 1 year post last islet transplantation. Additional follow-up may be provided at least annually for up to 9 years post first transplantation.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have had Type 1 diabetes mellitus for more than 5 years, and are exhibiting 1 of the following, despite intensive insulin management efforts: a) hypoglycemic unawareness, as defined by inability to sense hypoglycemia until the blood glucose falls to less than 54 mg/dL; b) metabolic instability, with 2 or more episodes of severe hypoglycemia (defined as an event with symptoms consistent with hypoglycemia in which the patient requires the assistance of another person and which is associated with a blood glucose below 54 mg/dL) or 2 or more hospital visits for diabetic ketoacidosis over the last year; or c) despite efforts at optimal glucose control, progressive secondary complications of diabetes as defined by retinopathy, nephropathy, or neuropathy.
* Are 18 to 65 years of age.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have had severe cardiac disease as defined by: a) recent myocardial infarction within the past 6 months; b) angiographic evidence of non-correctable coronary artery disease; or c) evidence of ischemia on a functional cardiac exam.
* Actively abuse alcohol or substances, including cigarette smoking (must not have smoked within the last 6 months).
* Have psychiatric problems that prevent them from being a suitable candidate for transplantation (such as schizophrenia, bipolar disorder, or major depression that is not controlled or stable on current medication).
* Have a history of not following prescribed regimens.
* Have active infection including hepatitis C virus, hepatitis B virus, human immunodeficiency virus (HIV), or Tuberculosis (TB) (or under treatment for suspected TB).
* Have a history of malignancy, except squamous or basal skin cancer.
* Weigh more than 70 kilograms or have a Body Mass Index (BMI) greater than 26 kg/m^2 at time of screening.
* Have a C-peptide value of 0.3 ng/ml or more following a 5.0 gram intravenous arginine infusion challenge.
* Are unable to provide informed consent.
* Have gallstones or hemangioma in liver.
* Have untreated proliferative retinopathy.
* Are breast-feeding or pregnant, or intend to try and become pregnant (females) or to father a child (males), or fail to follow birth control methods.
* Have had a previous transplant, or evidence of anti-human leukocyte antigen (HLA) antibody.
* Have an insulin requirement of more that 0.7 International Units (IU)/kilograms/day.
* Have a blood glycosylated hemoglobin (HbA1c) higher than 12 percent.
* Are unable to reach the hospital for transplantation within 2 hours of notification.
* Have untreated or treated hyperlipidemia.
* Have a medical condition requiring chronic use of steroids.
* Use coumadin or other anticoagulants (aspirin is allowed).
* Have Addison's disease.
* Have a negative screen for Epstein-Barr virus (EBV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2001-04; Primary Completion 2005-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (9):
- United States (5):
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Benaroya Research Institute at Virginia Mason Research Center, Seattle, Washington
- University of Alberta, Edmonton, Alberta, Canada
- Justus-Leibig University, Giessen, Germany
- University of Milan, Milan, Italy
- University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided to the public in : 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) portal.

REFERENCES:
- [Result] Shapiro AM, Ricordi C, Hering BJ, Auchincloss H, Lindblad R, Robertson RP, Secchi A, Brendel MD, Berney T, Brennan DC, Cagliero E, Alejandro R, Ryan EA, DiMercurio B, Morel P, Polonsky KS, Reems JA, Bretzel RG, Bertuzzi F, Froud T, Kandaswamy R, Sutherland DE, Eisenbarth G, Segal M, Preiksaitis J, Korbutt GS, Barton FB, Viviano L, Seyfert-Margolis V, Bluestone J, Lakey JR. International trial of the Edmonton protocol for islet transplantation. N Engl J Med. 2006 Sep 28;355(13):1318-30. doi: 10.1056/NEJMoa061267. PMID 17005949
- [Result] Brennan DC, Shannon MB, Koch MJ, Polonsky KS, Desai N, Shapiro J. Portal vein thrombosis complicating islet transplantation in a recipient with the Factor V Leiden mutation. Transplantation. 2004 Jul 15;78(1):172-3. doi: 10.1097/01.tp.0000128332.71657.ea. No abstract available. PMID 15257060
- [Derived] Benedini S, Ermetici F, Briganti S, Codella R, Terruzzi I, Maffi P, Caldara R, Secchi A, Nano R, Piemonti L, Alejandro R, Ricordi C, Luzi L. Insulin-mimetic effects of short-term rapamycin in type 1 diabetic patients prior to islet transplantation. Acta Diabetol. 2018 Jul;55(7):715-722. doi: 10.1007/s00592-018-1141-z. Epub 2018 Apr 13. PMID 29654388
- [Derived] Gala-Lopez B, Kin T, O'Gorman D, Pepper AR, Senior P, Humar A, Shapiro AM. Microbial contamination of clinical islet transplant preparations is associated with very low risk of infection. Diabetes Technol Ther. 2013 Apr;15(4):323-7. doi: 10.1089/dia.2012.0297. Epub 2013 Feb 25. PMID 23438305
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY567 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY567 — ImmPort study identifier is SDY567. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts and is available to the Public.
- Available data/document: Study summary, -schematic, -design, -adverse event(s),-medications,-demographics, - lab tests, -study files: SDY567 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY567 — ImmPort study identifier is SDY567. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts and is available to the Public.
- Available data/document: Individual Participant Data Set: ITN005CT — http://www.itntrialshare.org/project/Studies/ITN005CTPUBLIC/Study%20Data/begin.view? — TrialShare is the Immune Tolerance Network (ITN) portal that makes data from the consortium's clinical trials publicly available without charge. Creating an account for ITN TrialShare is free and allows for searching studies of interest.
- Available data/document: Study overview & protocol synopsis, -navigator, -schedule of assessments, -data&reports, -specimens, etc.: ITN005CT — http://www.itntrialshare.org/project/Studies/ITN005CTPUBLIC/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine centers recruited participants 18 to 65 years of age who had Type 1 diabetes mellitus for more than five years, recurrent neuroglycopenia that included reduced awareness of their hypoglycemic episodes or severe glycemic lability, and fulfilled all eligibility criteria. Refer to the Eligibility section for more details.
Groups:
- Islet Transplantation: Participants received portal vein islet infusions (up to 3), e.g., islet transplantations, with a targeted total of exceeding 10,000 islet equivalents per kilogram of body weight (IE/kg) per infusion. 25 participants received 2 transplantations and 16 participants received 3 transplantations. Participants received steroid-free post-transplantation immunosuppressive medications:
  1. Daclizumab 1 mg/kg intravenously immediately pre-transplantation and 2, 4, 6, and 8 weeks post-transplantation.
  2. Sirolimus 0.2 mg/kg by mouth once pre-transplantation then 0.1 mg/kg daily post-transplantation. Dosing was adjusted to achieve a trough peripheral blood level of 12-15 ng/mL x3 months after transplantation and 7-12 ng/mL for the remainder of the study.
  3. Tacrolimus 1 mg by mouth x1 pre-transplantation followed by 1 mg twice daily post transplantation. Levels were adjusted to achieve a peripheral blood trough level of 3-6 ng/mL for maintenance immunosuppression.
Period: Overall Study
Arm/Group | Islet Transplantation
Started | 36
Completed | 25 (One subject experienced pneumonia, myocardial infarction, and acute renal failure)
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 6
Not completed — Unknown Reasons | 2
Not completed — Immunosuppression-related Side Effects | 1

BASELINE CHARACTERISTICS:
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 22
Race/Ethnicity, Customized [Number; unit: Participants] — Race/Ethnicity (Reference: Public Health Service [PHS] 398/2590, Revised 6/2009)
  Participants
    Race: White | 35
    Race: Unspecified | 1
    Ethnicity: Non-Hispanic | 36
Region of Enrollment [Number; unit: participants]
  United States | 19
  Canada | 4
  Germany | 4
  Italy | 4
  Switzerland | 5
Number of Years with Diabetes [Mean (Standard Deviation); unit: Years] — Average number of years at baseline visit since the participant was physician-diagnosed with Type 1 diabetes mellitus (T1DM)
  Years | 27 (10.4)
Daily Insulin Usage [Mean (Standard Deviation); unit: Units of Insulin/kilogram/day (U/kg/day)] — Average daily insulin usage at baseline visit
  Units of Insulin/kilogram/day (U/kg/day) | 0.5 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants That Achieved Insulin Independence With Adequate Control of Blood Glucose Levels at One Year Post Final Islet Transplantation.
Description: Insulin independence: exogenous insulin not required and glycemic control is achieved as defined by maintaining 1.) a blood glycosylated hemoglobin (HbA1c) level < 6.5% (Normal:<5.7%; pre-diabetes: 5.7% -6.4%; diabetes: 6.5% or higher),2) a blood glucose level after an overnight fast not exceeding 140 mg per deciliter (dL) more than three times in any week (Normal: 70 to 120 mg/dL), and 3)not exceeding a 2-hour postprandial blood glucose level of 180 mg/dL more than four times per week (Normal: <140mg/dL if <=50 years of age, <150 mg/dL for ages 50-60 years and <160 mg/dL for ages 60+)
Time Frame: One year status post participant receipt of final islet transplantation
Population: Intent-to-treat
Measure: Number; unit: Percent of Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 36
Percent of Participants
  Insulin Independence at One Year | 44
  Insulin Independence with One Transplant | 14
  Insulin Independence with Two Transplants | 17
  Insulin Independence with Three Transplants | 14
Statistical Analysis 1: Comparison: Islet Transplantation; Test type: Superiority or Other; Fisher Exact; Odds Ratio (OR) = 44, 95% CI 2-sided [30 to 61]

2. Secondary Outcome: Percent of Participants With Partial Islet Function One Year Post Final Islet Transplantation.
Description: Partial islet function definition: a fasting basal C-peptide level >= 0.3 ng/mL and a continuing need for insulin or suboptimal glycemic control (Note: C-peptide is a substance that the pancreas releases into the bloodstream in equal amounts to insulin, thereby showing how much insulin the body is making). Adequate glycemic control is defined by: 1) a blood HbA1c level <6.5%, 2) a blood glucose level after an overnight fast not exceeding 140 mg/dL more than three times in any week and, 3) a 2-hour postprandial blood glucose level not exceeding 180 mg/dL more than four times per week
Time Frame: One year post receipt of final islet transplantation
Population: Intent-to-treat
Measure: Number; unit: Percent of Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 36
Percent of Participants | 28
Statistical Analysis 1: Comparison: Islet Transplantation; Test type: Superiority or Other; Fisher Exact; Odds Ratio (OR) = 28, 95% CI 2-sided [16 to 44]

3. Secondary Outcome: Percent of Participants That Achieved Insulin Independence From First Transplant
Description: Insulin independence: exogenous insulin not required and glycemic control is achieved as defined by maintaining 1) a blood glycosylated hemoglobin (HbA1c) level < 6.5% (Normal:<5.7%; pre-diabetes: 5.7% -6.4%; diabetes: 6.5% or higher),2) a blood glucose level after an overnight fast not exceeding 140 mg per deciliter (dL) more than three times in any week (Normal: 70 to 120 mg/dL), and 3)not exceeding a 2-hour postprandial blood glucose level of 180 mg/dL more than four times per week (Normal: <140mg/dL if <=50 years of age, <150 mg/dL for ages 50-60 years and <160 mg/dL for ages 60+)
Time Frame: First transplantation until end of study (up to six years post final transplantation)
Population: Intent-to-Treat
Measure: Number; unit: Percent of Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 36
Percent of Participants | 58
Statistical Analysis 1: Comparison: Islet Transplantation; Test type: Superiority or Other; Fisher Exact; Odds Ratio (OR) = 58, 95% CI 2-sided [42 to 63]

4. Secondary Outcome: Percent of Participants With Detectable Fasting Basal C-Peptide Levels
Description: C-peptide is a substance that the pancreas releases into the bloodstream in equal amounts to insulin, thereby showing how much insulin the body is making. C-peptide secretion is used to measure the function of transplanted islets. Higher levels indicate better islet function. Detectable fasting basal levels of C-peptide secretion are >=0.3 ng/ml.
Time Frame: Two years post first transplantation
Population: Intent-to-Treat
Measure: Number; unit: Percent of Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 36
Percent of Participants | 70

5. Post Hoc Outcome: HbA1c Plasma Laboratory Values for Participants in the Extended Follow-up Study Phase
Description: Seven participants from US sites were included in the extended follow-up. These participants were monitored yearly from year three post last transplantation (the original end of study follow-up) through August 30, 2010 (up to 9 years post first transplantation), at which point they were transferred to a new protocol (ITN040CT [NCT01309022]). Glycosylated hemoglobin (HbA1c) is a measure of the average plasma glucose concentration over prolonged periods of time. (Normal:<5.7%; pre-diabetes: 5.7% -6.4%; diabetes: 6.5% or higher)
Time Frame: First transplantation through August 30, 2010 (up to 9 years)
Population: Intent-to-Treat
Measure: Mean (Full Range); unit: HbA1c Percentage
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 7
HbA1c Percentage | 6.2 [6.0 to 6.5]

6. Post Hoc Outcome: Serum Creatinine Levels for Participants in the Extended Follow-up Study Phase
Description: Seven participants from US sites were included in the extended follow-up. These participants were monitored yearly from year three post last transplantation (the original end of study follow-up) through August 30, 2010 (up to 9 years post first transplantation), at which point they were transferred to a new protocol (ITN040CT [NCT01309022]). Serum creatinine is a measure of renal function. Normal ranges are from 0.5 to 1.0 mg/dL for females and 0.7 to 1.2 mg/dL for males.
Time Frame: First transplantation through August 30, 2010 (up to 9 years)
Population: Intent-to-Treat
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 7
mg/dL | 0.9 [0.7 to 1.6]

ADVERSE EVENTS:
Time Frame: First transplant until end of study (up to 9 years post first transplant)
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Toxicity Criteria Version 2.0 (April 30, 1999)
Arm/Group | Islet Transplantation
Serious Adverse Events (participants affected / at risk) | 17/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Myocardial infarction (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (3)
Appendiceal abscess (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2)
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatic haemangioma rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation (N=36)
Anaemia (Blood and lymphatic system disorders) | 29 (133)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 27 (119)
Lymphopenia (Blood and lymphatic system disorders) | 9 (30)
Neutropenia (Blood and lymphatic system disorders) | 19 (114)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (43)
Bradycardia (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 3 (4)
Pericardial effusion (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vision blurred (Eye disorders) | 3 (4)
Vitreous floaters (Eye disorders) | 3 (3)
Vitreous haemorrhage (Eye disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 12 (20)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13)
Aphthous stomatitis (Gastrointestinal disorders) | 4 (6)
Constipation (Gastrointestinal disorders) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 23 (52)
Dyspepsia (Gastrointestinal disorders) | 4 (8)
Flatulence (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Lip ulceration (Gastrointestinal disorders) | 2 (2)
Loose stools (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 33 (138)
Nausea (Gastrointestinal disorders) | 19 (28)
Tongue ulceration (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 15 (31)
Asthenia (General disorders) | 5 (8)
Chest discomfort (General disorders) | 2 (2)
Chest pain (General disorders) | 2 (5)
Fatigue (General disorders) | 14 (24)
Influenza like illness (General disorders) | 3 (4)
Malaise (General disorders) | 2 (3)
Mucosal ulceration (General disorders) | 3 (4)
Oedema (General disorders) | 6 (6)
Oedema peripheral (General disorders) | 9 (13)
Pain (General disorders) | 6 (8)
Pyrexia (General disorders) | 11 (15)
Rigors (General disorders) | 3 (4)
Portal hypertension (Hepatobiliary disorders) | 4 (4)
Hypersensitivity (Immune system disorders) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3)
Cellulitis (Infections and infestations) | 3 (3)
Clostridium colitis (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 4 (4)
Fungal infection (Infections and infestations) | 3 (7)
Herpes simplex (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Hordeolum (Infections and infestations) | 2 (4)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 11 (12)
Onychomycosis (Infections and infestations) | 4 (4)
Rhinitis (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 4 (4)
Tonsillitis (Infections and infestations) | 2 (3)
Tooth abscess (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 8 (10)
Urinary tract infection (Infections and infestations) | 9 (13)
Vaginal candidiasis (Infections and infestations) | 2 (2)
Vaginal mycosis (Infections and infestations) | 4 (6)
Viral infection (Infections and infestations) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (4)
Excoriation (Injury, poisoning and procedural complications) | 3 (3)
Incision site complication (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 9 (14)
Aspartate aminotransferase increased (Investigations) | 10 (17)
Band neutrophil percentage increased (Investigations) | 2 (2)
Blood albumin decreased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (4)
Blood bicarbonate decreased (Investigations) | 5 (18)
Blood chloride increased (Investigations) | 2 (9)
Blood cholesterol increased (Investigations) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Blood urea increased (Investigations) | 3 (3)
Hepatic enzyme increased (Investigations) | 12 (20)
Liver function test abnormal (Investigations) | 14 (20)
Mean cell volume decreased (Investigations) | 3 (4)
Red blood cell count decreased (Investigations) | 5 (14)
Weight decreased (Investigations) | 9 (11)
White blood cell count decreased (Investigations) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5)
Hyperchloraemia (Metabolism and nutrition disorders) | 3 (6)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 (18)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 (9)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (8)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (9)
Hypoglycaemia (Metabolism and nutrition disorders) | 11 (24)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (25)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (6)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 6 (9)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Amnesia (Nervous system disorders) | 2 (2)
Burning sensation (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 20 (53)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 3 (4)
Migraine (Nervous system disorders) | 4 (4)
Paraesthesia (Nervous system disorders) | 3 (4)
Tremor (Nervous system disorders) | 9 (13)
Anxiety (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 6 (8)
Nocturia (Renal and urinary disorders) | 2 (4)
Proteinuria (Renal and urinary disorders) | 3 (6)
Renal cyst (Renal and urinary disorders) | 2 (2)
Menstrual disorder (Reproductive system and breast disorders) | 2 (2)
Menstruation irregular (Reproductive system and breast disorders) | 5 (7)
Ovarian cyst (Reproductive system and breast disorders) | 3 (7)
Vaginal discharge (Reproductive system and breast disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (19)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 15 (25)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (7)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 3 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (10)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 13 (18)
Rash papular (Skin and subcutaneous tissue disorders) | 3 (6)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (4)
Haematoma (Vascular disorders) | 4 (5)
Hot flush (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 7 (11)
Hypotension (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No